CLINICAL TRIAL: NCT02028156
Title: Evaluation of Feeding Intolerance in Formula-Fed Infants: A Non-Randomized, Single-Group, Multi-Center Study
Brief Title: Feeding Intolerance in Formula-Fed Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DA06
Record Dates: First submitted 2013-12-06; First posted 2014-01-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Feeding Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Partially Hydrolyzed Infant Formula (Experimental): Fed ad lib.
  Interventions: Other: Partially Hydrolyzed Infant Formula

INTERVENTIONS:
Other: Partially Hydrolyzed Infant Formula — Commercially available infant formula

SUMMARY:
This is a non-randomized, single-group, multi-center, two phased study to evaluate formula intolerance.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Stage 1:

* Singleton full term birth with birth weight of > 2500g.
* Infant between 0 and 60 days of age.
* Discontinuation of medications that might affect gastrointestinal (GI) tolerance.
* Infant is exclusively formula-fed a full-lactose, intact cow milk protein-based infant formula (CMF) for less than 7 days prior to enrollment.

Inclusion Criteria for Stage 2:

* Infant was fed according to protocol in Stage 1 of the study.
* Infant was identified as being fussy using the Intolerance Assessment Tool in Stage 1.

Exclusion Criteria:

Exclusion Criteria for Stage 1:

* Chromosomal or major congenital anomalies.
* Suspected or known metabolic or physical diseases affecting infant feeding and/or metabolism.
* Hospitalization, other than for delivery, prior to enrollment.
* Severe uncontrolled eczema, visible bloody stools or milk protein allergy prior to enrollment.
* More than 1 substitution of an infant formula other than full-lactose, intact cow milk formula (CMF) since birth.
* Use of a prokinetic drug within 7 days before enrollment.

Exclusion Criteria for Stage 2:

* Infant's intolerance symptom was caused by another reason, for example known infection/illness, food allergy, or response to vaccination(s).
* Infant has immunization(s) within 3 days of enrollment in Stage 2.

Max Age: 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Improvement in Fussiness | 0 to 15 days
  Study phase 2; Parent completed questionnaire.

SECONDARY OUTCOMES:
Diarrhea | 0 to 4 weeks
  Study phase 1; Parent completed questionnaire.
Constipation | 0 to 4 weeks
  Study phase 1; Parent completed questionnaire.
Spit-up | 0 to 4 weeks
  Study phase 1; Parent completed questionnaire.
Gassiness | 0 to 4 weeks
  Study phase 1; Parent completed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Li, MD, Study Chair — Abbott Nutrition China
Locations (3):
- China (3):
  - Guangdong Women and Children Hospital, Guangzhou, Guangdong
  - Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - Xin Hua Hospital, Shanghai